CLINICAL TRIAL: NCT03431935
Title: Longitudinal Examination of Predictors and Outcomes of Sickle Cell Disease Healthcare Transition
Brief Title: Predictors and Outcomes in Patients With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Methodist Comprehensive Sickle Cell Center (Unknown); University of Memphis (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LEAPS; K01HL125495-01A1 (NIH)
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Disease
Keywords: Health Care Transition; Adolescent; Young Adult
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Children with sickle cell disease (SCD) are living longer with the advent of medical advances such as prophylactic penicillin, chronic transfusion, and hydroxyurea. Despite greater longevity in SCD, the period following the transition from pediatric to adult care is critical; youth aged 18-30 years are at high risk for mortality and have high rates of healthcare utilization, leading to high healthcare costs. As such, health care transition (HCT) programs have been created to prepare patients for adult-centered care and subsequently, improve health outcomes. However, very few programs have been evaluated for effectiveness in achieving optimal health outcomes in SCD. This paucity of program evaluation is attributed to a lack of identifiable predictors and outcomes.

Researchers at St. Jude Children's Research Hospital want to identify factors and patterns of successful HCT. This information will be used to develop approaches to best evaluate HCT interventions and identify areas of improvement of HCT programming.

PRIMARY OBJECTIVE: Describe hospital utilization, treatment adherence, and health-related quality of life in a cohort of patients with sickle cell disease (SCD) who will transfer to adult care during the study period.

SECONDARY OBJECTIVE: Examine the associations between various factors and health care transition (HCT) outcomes.

DETAILED DESCRIPTION:
Participants will be asked to complete a set of questions during an outpatient clinic visit at St. Jude or Methodist Adult Comprehensive Sickle Cell Center. The questions ask about sickle cell disease knowledge and self-management skills, access to care, general adjustment, quality of life, and stress. These questions will take about 60 minutes to complete.

Participants will answer questionnaires on a password protected laptop or tablet using a computer program called Audio Computer-Assisted Self-Interviews (ACASI). The laptop or tablet will be kept by the study team. A study team member will be available during this time to address any technical issues or answer any questions. Participants will answer one of the questionnaires verbally, and the study team member will record responses from the questionnaire with paper and pen. Questionnaires given verbally will be audio-recorded and reviewed by the lead researcher or other study team member. The recordings will be destroyed immediately after review. No transcript or written record of the recordings will be made. Study members will meet five times with each participant during regularly-scheduled clinical visits over a two year period.

Two institutions will collaborate in the proposed project. St. Jude Children's Research Hospital (St. Jude) and the Methodist Comprehensive Sickle Cell Center will be the primary source of participants. Faculty from the University of Memphis, Department of Psychology, will be involved in methodological considerations and analyzing the data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell disease (all genotypes).
* Age 16.0 - 20.99 years at initial assessment.
* Primary language is English.

Exclusion Criteria:

* Participant unable to complete the questionnaires due to refusal, current acute illness (e.g., pain crisis), or significant cognitive impairment as judged by health care providers at the SCD clinic.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants who meet eligibility criteria and have a pre-existing relationship as a patient at St. Jude Children's Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Number of emergency room/hospital admissions in the previous 12 months | Once, at age 19
  The primary objective will utilize data collected at age 19 years, 0 months (±2 months), the age participants will have transferred to adult care. This data will come from participants enrolled between the ages of 17 years, 0 months and 19 years, 0 months.
Percent of clinic visits completed in the previous 12 months | Once, at age 19
  The primary objective will utilize data collected at age 19 years, 0 months (±2 months), the age participants will have transferred to adult care. This data will come from participants enrolled between the ages of 17 years, 0 months and 19 years, 0 months.
Percent hydroxyurea prescription refill rate | Once, at age 19
  The primary objective will utilize data collected at age 19 years, 0 months (±2 months), the age participants will have transferred to adult care. This data will come from participants enrolled between the ages of 17 years, 0 months and 19 years, 0 months.
Health-related quality of life as assessed by the PedsQL | Once, at age 19
  The primary objective will utilize data collected at age 19 years, 0 months (±2 months), the age participants will have transferred to adult care. This data will come from participants enrolled between the ages of 17 years, 0 months and 19 years, 0 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jerlym Porter, PhD, MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - Methodist Adult Comprehensive Sickle Cell Center, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org
- See also: Methodist Comprehensive Sickle Cell Center — http://www.methodisthealth.org/healthcare-services/sickle-cell-center/